CLINICAL TRIAL: NCT03909438
Title: Investigation and Study on the Status of Endovascular Therapy in Acute Ischemic Stroke
Brief Title: Investigation and Study on the Status of Endovascular Therapy in Acute Ischemic Stroke Ischemic Stroke
Acronym: IS-EVT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Fourth Affiliated Hospital, School of Medicine, Zhejiang University (Unknown); Taizhou Hospital (Other); Lishui Country People's Hospital (Other); The Central Hospital of Lishui City (Other); Shaoxing People's Hospital (Other); Ganzhou People's Hospital (Unknown); Luoyang Central Hospital (Other); Huizhou Municipal Central Hospital (Other); The Second Affiliated Hospital of Jiaxing University (Other); Shanghai Zhongshan Hospital (Other); The First People's Hospital of Huzhou (Other); Taizhou First People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IS-EVT
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Stroke; Endovascular Therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endovascular Thrombectomy — Endovascular therapy includes direct mechanical thrombectomy or intravenous thrombolysis with mechanical thrombectomy. Endovascular Thrombectomy Device: Trepo trevor Retriever Device: SolitaireTM FR Revascularization Device

SUMMARY:
This study aims to build a database for patients with acute ischemic stroke who receive endovascular therapy and analyze the current situation, effectiveness, safety and cost-effectiveness of endovascular therapy for acute ischemic stroke in China.

DETAILED DESCRIPTION:
Study design is a registry, prospective, multicenter study of acute ischemic stroke patients with endovascular treatment. A database will be established including age, gender, smoking history, blood pressure, blood glucose, previous history (such as coronary heart disease, atrial fibrillation, hypertension, diabetes, stroke history, etc.), history of antiplatelet drugs, onset to treatment time, National Institute of Health Stroke Scale (NIHSS) score before treatment.

Indications for endovascular therapy refer to the current guidelines. All patients will receive endovascular therapy, including direct endovascular therapy or intravenous thrombolysis with endovascular therapy. The effectiveness, safety and cost-effectiveness of endovascular therapy for acute ischemic stroke will be analyzed.

This study will enroll up at least 1,000 patients in 70 centers in China. The primary end point are proportion of patients with good prognosis after 90 days and intracranial hemorrhage transformation type after 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical signs and symptoms consistent with the diagnosis of an acute ischemic stroke
2. Age ≥18 years
3. NIHSS ≥ 6
4. ICA or MCA-M1 or MCA-M2 occlusion as evidenced by MRA or 4D-CTA
5. Ethrombectomy can be initiated (femoral puncture) within 6 hours after onset or between 6 and 24 hours after time last know well if conform to the imaging inclusion criteria: Target Mismatch Profile on CT perfusion or MR perfusion: ischemic core volume is ≤ 70 ml, mismatch ratio is ≥ 1.8, penumbra volume is ≥ 15 ml.

Exclusion Criteria:

1. Large area cerebral infarction of anterior circulation on early CT image (more than 1/3 of cerebral hemisphere)
2. Blood glucose <2.7mmol/L or >22.2mmol/L
3. Other serious, advanced, or terminal illness (investigator judgment) or life expectancy is less than 90 days
4. Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients will receive endovascular therapy, including direct endovascular therapy or intravenous thrombolysis with endovascular therapy.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Good Functional Independence | 90 days
  This outcome will look at the proportion of patients with mRS 0-2 at day 90.
Hemorrhage transformation | 24-hour
  hemorrhage transformation at 24-hour after reperfusion therapy:
  * Hemorrhagic infarction 1 (HI1) was defined as small petechiae along the margins of the infarct;
  * Hemorrhagic infarction 2 (HI2) as confluent petechiae within the infarcted area but no space-occupying effect;
  * Parenchymal hemorrhage (PH1) as blood clots in 30% or less of the infarcted area with some slight space- occupying effect; and
  * Parenchymal hemorrhage (PH2) as blood clots in more than 30% of the infarcted area with substantial space- occupying effect.
  * Symptomatic intracranial hemorrhage was defined as blood at any site in the brain on the CT scan.

SECONDARY OUTCOMES:
Poor outcome | 90 days
  This outcome will look at the proportion of patients with mRS 3-6 at day 90.
The incidence of recurrent stroke or other vascular events | 90 days
  The incidence of recurrent stroke and other vascular events at 90 days after endovascular therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Min Lou, Ph.D, Study Director — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided